CLINICAL TRIAL: NCT05702632
Title: Comparison of Thera-togs Orthotics With Reciprocal Electrotherapy for Postural Stability in Spastic Diplegic Cerebral Palsy
Brief Title: TheraTogs Versus Reciprocal Electrical Stimulation on Children With Diplegic Cerebral Palsy: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Reffat, lecturer at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Approaches
Record Dates: First submitted 2022-10-27; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Device: 1- Reciprocal electrical stimulation; Procedure: traditional physical therapy program
- Group B (Active Comparator)
  Interventions: Device: TheraTogs orthotic treatment; Procedure: traditional physical therapy program

INTERVENTIONS:
Device: 1- Reciprocal electrical stimulation — A specialized programmable electrical stimulation device was used (Uniphy is the manufacturer of Phyaction787; Uniphy, Eindhoven, the Netherlands). The device has two channels that can alternatively stimulate two opposing groups of muscles (reciprocate).
  Arms: Group A
Device: TheraTogs orthotic treatment — A sleeveless top vest and two pairs of shorts with two thigh cuffs and limb cuffs each make up the TheraTogs strapping system which is applied to the children in the TheraTogs group. The TheraTogs suit is providing breathable, comfortable- Latex over the torso and thigh, as well as free toileting. For infection control and size fitting problems, participants are not allowed to share their TheraTogs with other patients. TheraTog's orthotic undergarment and strapping system were worn under their regular clothes, so it was neither distracting nor irritating.
  Arms: Group B
Procedure: traditional physical therapy program — Facilitation of balance and gait training

SUMMARY:
Children with diplegic cerebral palsy exhibit postural restrictions as a result of both primary and secondary brain damage impairments. One of the main goals of cerebral palsy rehabilitation is to improve balance and stability. As a result, the purpose of this study is to compare the effects of TheraTogs and reciprocal electrical stimulation on postural stability in children with diplegic CP.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic children of both sexes are between the ages of 8 and 12. The level of spasticity in the lower limbs ranged from grade 1 to grade +1 on the modified Ashworth scale (MAS). The levels of motor function were between levels I and II, according to the Gross Motor Function Classification System (GMFCS).

Exclusion Criteria:

* If they had no major medical issues, according to their medical report. Skin diseases and allergic reactions to the adhesive tape used in this study were excluded, as were any deformities that interfered with lower limb functions, children with pace- makers who were contraindicated by electrical stimula- tion, children with visual, auditory, or perceptual deficits, and children with seizures.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
postural stability | 3 months
  overall stability indices had been measured by Biodex balance system

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Eldoky, Egypt